CLINICAL TRIAL: NCT06600022
Title: A Phase I/II, Open-label, Multicentre, Dose-escalation, and Dose-expansion Study to Evaluate the Safety, Pharmacokinetics and Anti-tumor Activity of SCTB41 in Patients with Advanced Malignant Solid Tumours
Brief Title: Aims to Explore the Safety, Tolerability, and Preliminary Efficacy of SCTB41 in Adult Patients with Advanced Malignant Solid Tumours.
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCTB41-X101
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10

CONDITIONS: Advanced Malignant Solid Tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arms (Experimental): SCTB41 of different doses,IV,every 3 weeks
  Interventions: Drug: SCTB41

INTERVENTIONS:
Drug: SCTB41 — SCTB41 of different doses,IV,every 3 weeks

SUMMARY:
This study aims to explore the safety, tolerability, PK characteristics, immunogenicity, and preliminary anti-tumor efficacy of SCTB41 as a monotherapy in adult patients with advanced malignant solid tumours. This study is an open label, multicentre, dose-escalation and dose-expansion Phase I/II clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form (ICF);
2. Male or female, ≥18 years old;
3. Survival duration more than 3 months;
4. ECOG score ≤ 1 point;
5. Participants in Phase Ia (dose-escalation phase) are required to meet the following criteria: histologically or cytologically confirmed diagnosis of advanced malignant solid tumour;
6. Participants in Phase Ib (dose-expansion phase) and Phase II are required to meet the following criteria: Histologically or cytologically confirmed specific type advanced malignant solid tumours;
7. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Participants with brainstem, meningeal, spinal metastases, orcompression; active central nervous system metastases;
2. Other malignancies diagnosed;
3. History of hypertensive crisis or hypertensive encephalopathy; presence of uncontrolled hypertension. History of arterial thrombosis or deep veinthrombosis within 6 months prior to enrollment;
4. Presence of any active autoimmune disease or a history of autoimmunedisease with an expected recurrence;
5. Received chemotherapy, immunotherapy, biologic therapy, or other antitumor treatments within 4 weeks before enrollment;
6. Need for immunosuppressive drugs within 2 weeks prior to enrollment oranticipated during the study;
7. Significant coagulopathy or other evident risk of bleeding;
8. uncontrolled effusions in the serous cavities within 4 weeks before enrollment；
9. Major surgery or significant trauma within 4 weeks prior to enrollment;presence of unhealed skin wounds, surgical sites, trauma sites, severe- Page 3 of 4 [DRAFT] -mucosal ulcers, or fractures, or if the Investigator deems the participantunsuitable for the study;
10. History of permanent discontinuation of immunotherapy due to immunerelated toxicity or occurrence of ≥ Grade 3 irAEs;
11. Known severe allergy to similar antibody drugs;
12. Presence of active infection；
13. History of organ transplantation or stem cell transplantation;
14. Pregnant or breastfeeding female; women of childbearing potential withpositive pregnancy test within 7 days before the enrollment; participants(including males of childbearing potential and their female partners, and females of childbearing potential and their male partners) unwilling to use medically recognized effective contraception during the study and for 6 months after treatment ends.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting toxicity(DLT) | :From Day 0 up to Day 21
  Incidence of dose-limiting toxicities up to the Day 21 visit
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with SCTB41 until the first documentation ofdisease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with SCTB41 until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China